CLINICAL TRIAL: NCT00683384
Title: A Prospective, Observational Study to Monitor Safety in Patients Who Were Administered With Etanercept (Enbrel) 25 mg by Subcutaneous Injection
Brief Title: Study Evaluating the Safety of Enbrel (Etanercept)
Status: Completed | Type: Observational
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Other Study IDs: 0881A-102300
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Results first posted 2010-11-16 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-10

CONDITIONS: Arthritis, Psoriatic
Keywords: Arthritis; psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic; Arthritis | interventions — Etanercept

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Drug: Etanercept (Enbrel)

INTERVENTIONS:
Drug: Etanercept (Enbrel)

SUMMARY:
The purpose of this study is to collect post-marketing information on the safety of Enbrel in Filipino patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients from the study center who received or will receive at least one dose of Enbrel according to the approved product indication.

Exclusion Criteria:

* Previously discontinued Enbrel therapy due to significant safety concern.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2007-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Metro Manila, Philippines

RESULTS

PARTICIPANT FLOW:
Groups:
- Etanercept: Etanercept (Enbrel) 25 mg by subcutaneous injection
Period: Overall Study
Arm/Group | Etanercept
Started | 93
Completed | 91
Not Completed | 2
Not completed — Death | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Etanercept
Number analyzed (Participants) | 93
Age Continuous [Mean (Standard Deviation); unit: years] | 41.8 (18.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 45

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Spontaneous Adverse Events Reported Until 30 Days After Each Injection
Time Frame: 30 days post injection up to 3 years
Population: Full analysis set
Measure: Number; unit: Participants
Arm/Group | Etanercept
Number analyzed (Participants) | 93
Participants | 7

ADVERSE EVENTS:
Arm/Group | Etanercept
Serious Adverse Events (participants affected / at risk) | 1/93
Other Adverse Events (participants affected / at risk) | 6/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=93)
Death (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=93)
Hyperhidrosis (General disorders) | 1
Injection site irritation (General disorders) | 1
Injection site pruritus (General disorders) | 1
Transaminases increased (Investigations) | 1
Formication (Nervous system disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.